CLINICAL TRIAL: NCT05275010
Title: A Randomized, Open-Label, 2-Arm, Parallel Group, Single Dose, Multi-Centre Study in Healthy Male Subjects to Investigate the Comparability of Pharmacokinetics of the Fixed-Dose Combination of Pertuzumab and Trastuzumab Administered Subcutaneously Using a Handheld Syringe or Using the On-Body Delivery System
Brief Title: A Study in Healthy Male Subjects to Investigate the Comparability of Pharmacokinetics of the Fixed-Dose Combination of Pertuzumab and Trastuzumab Administered Subcutaneously Using a Handheld Syringe or Using the On-Body Delivery System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WP42873
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — pertuzumab; Trastuzumab; Needles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: PH FDC SC Using a Handheld Syringe (Active Comparator): A single dose of PH FDC SC (600 mg pertuzumab/600 mg trastuzumab) will be administered by a healthcare professional subcutaneously (SC) into the participant's anterior thigh on Day 1, using a handheld syringe with hypodermic needle.
  Interventions: Drug: Fixed-Dose Combination of Pertuzumab and Trastuzumab SC (PH FDC SC); Device: Handheld Syringe with Hypodermic Needle
- Arm 2: PH FDC SC Using the OBDS (Experimental): A single dose of PH FDC SC (600 mg pertuzumab/600 mg trastuzumab) will be administered by a healthcare professional subcutaneously (SC) into the participant's anterior thigh on Day 1, using the on-body delivery system (OBDS).
  Interventions: Drug: Fixed-Dose Combination of Pertuzumab and Trastuzumab SC (PH FDC SC); Device: On-Body Delivery System

INTERVENTIONS:
Drug: Fixed-Dose Combination of Pertuzumab and Trastuzumab SC (PH FDC SC) — A single dose of PH FDC SC (600 mg pertuzumab/600 mg trastuzumab) will be administered by a healthcare professional subcutaneously (SC) into the anterior thigh, using either a handheld syringe with hypodermic needle (Arm 1) or the on-body delivery system (Arm 2).
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; PHESGO®; RO7198574; RG6264
Device: Handheld Syringe with Hypodermic Needle — A single 10-mL dose of PH FDC SC will be administered as a subcutaneous (SC) injection using a handheld manual syringe.
  Arms: Arm 1: PH FDC SC Using a Handheld Syringe
Device: On-Body Delivery System — A single 10-mL dose of PH FDC SC will be administered as a subcutaneous (SC) injection using the on-body delivery system (OBDS).
  Arms: Arm 2: PH FDC SC Using the OBDS

SUMMARY:
This is a randomized, open-label, 2-arm, parallel-group, single-dose, multi-center study in healthy male subjects to investigate the comparability of the pharmacokinetics of the fixed-dose combination of pertuzumab and trastuzumab administered subcutaneously using the proprietary on-body delivery system or a handheld syringe with hypodermic needle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age 18-45 years at time of signing Informed Consent Form
* Ability to comply with the study protocol
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, during the treatment period and for 7 months after the dose of PH FDC SC
* A body mass index (BMI) between 18 and 32 kilograms per metre squared (kg/m2), inclusive
* Intact normal skin without potentially obscuring tattoos, pigmentation, or lesions in the area for intended injection on the thighs
* Baseline LVEF≥55% measured by echocardiogram (ECHO)
* No history of hypersensitivity or confirmed, clinically significant and clinically relevant allergic reactions, either spontaneously or following any drug administration
* No history of any clinically significant and clinically relevant cardiac condition
* No history of previous anticancer treatments including pertuzumab, trastuzumab, anthracyclines, or any cardiotoxic drugs
* No apparent family history of clinically significant and clinically relevant hypersensitivity, allergy, and severe cardiac diseases
* No contraindications from detailed medical and surgical history and physical examinations
* No previous enrollment in this study protocol and no concurrent enrollment in any other study protocol

Exclusion Criteria:

* Positive urine test for drugs of abuse as per local standard (for alcohol abuse, positive breath test is also acceptable)
* Positive test result for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) 1 or 2, showing: History of exposure to HBV, HCV, or HIV; or Active viral hepatitis infection (HBV or HCV) or HIV infection
* Systolic blood pressure ≥140 millimetres of mercury (mmHg) or <90 mmHg, or diastolic blood pressure >90 mmHg or <50 mmHg
* Use of prohibited medications including non-prescription medications, nutraceuticals, nutritional supplements or any herbal remedies taken within 10 days or 5 times the elimination half-life (whichever is longer) prior to randomization into the study
* Concomitant subcutaneous, intravenous, or any parenteral drugs within 90 days prior to screening
* Participation in an investigational drug or device study within 90 days or five times the elimination half-life (whichever is longer) prior to screening
* Donation of blood over 500 millilitres (mL) within 3 months prior to enrollment
* Known severe hypersensitivity to plaster, medical adhesive tapes, or bandages
* Known allergy to murine proteins, hyaluronidase, bee, or vespid venom, or any other ingredient in the formulation of rHuPH20 (Hylenex® recombinant [hyaluronidase human injection]) or any other ingredients and excipients in the formulation of PH FDC SC
* Clinically significant abnormalities in laboratory test results (including hepatic and renal panels, CBC, chemistry panel, and urinalysis)
* Clinically relevant electrocardiogram abnormalities at screening or Day -1
* History of any cardiac condition
* Lower extremity edema or pathology (e.g., cellulitis, lymphatic disorder or prior surgery, pre-existing pain syndrome, previous lymph node dissection etc.) that could interfere with any protocol-specified outcome assessment
* Any history of clinically significant and clinically relevant allergies, oncologic, psychiatric, gastrointestinal, renal, hepatic, cardiovascular or pulmonary disease
* Concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in this study
* Any clinically relevant history of systemic disease (e.g., malignancy, diabetes mellitus, gastrointestinal, renal, hepatic, cardiovascular, rheumatological, or pulmonary disease)
* History of breast cancer or treatment for breast cancer
* Current chronic daily treatment (continuous for >3 months) with corticosteroids (dose ≥10 mg/day methylprednisolone), excluding inhaled corticosteroids
* Receipt of intravenous antibiotics for infection within 7 days prior to enrollment into the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Australia (3):
  - Q-Pharm Pty Ltd; Nucleus Network Brisbane Clinic, Herston, Queensland
  - CMAX Pty Ltd, Adelaide, South Australia
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- New Zealand (2):
  - New Zealand Clinical Research - Auckland, Auckland
  - New Zealand Clinical Research - Christchurch, Christchurch

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Wynne C, Wang B, Deng R, Li J, Eiger D, Bene Tchaleu F, Heeson S, Restuccia E. Pharmacokinetic bioequivalence of the fixed-dose combination of pertuzumab and trastuzumab administered subcutaneously using a handheld syringe or an on-body delivery system. J Cancer Res Clin Oncol. 2025 Jun 14;151(6):188. doi: 10.1007/s00432-025-06228-4. PMID 40514611

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: PH FDC SC Using a Handheld Syringe: A single dose of PH FDC SC (600 mg pertuzumab/600 mg trastuzumab) was administered by a healthcare professional subcutaneously (SC) into the participant's anterior thigh on Day 1, using a handheld syringe with hypodermic needle.
- Arm 2: PH FDC SC Using the OBDS: A single dose of PH FDC SC (600 mg pertuzumab/600 mg trastuzumab) was administered by a healthcare professional subcutaneously (SC) into the participant's anterior thigh on Day 1, using the on-body delivery system (OBDS).
Period: Overall Study
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Started | 76 | 75
Received the Single Dose of Study Treatment (Safety Population) | 72 (4 participants discontinued the study prior to dosing on Day 1.) | 74 (1 participant discontinued the study prior to dosing on Day 1.)
Entered Follow-Up | 71 (1 participant withdrew from the study before follow-up.) | 74
Completed | 71 | 73 (1 participant was lost to follow-up.)
Not Completed | 5 | 2
Not completed — Reason Not Specified | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Median (Full Range); unit: Years] | 29.0 [18.0 to 46.0] | 29.0 [18.0 to 45.0] | 29.0 [18.0 to 46.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 76 | 75 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 68 | 65 | 133
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 15 | 13 | 28
  Native Hawaiian or Other Pacific Islander | 10 | 7 | 17
  Black or African American | 0 | 0 | 0
  White | 44 | 45 | 89
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 3 | 4 | 7
Number of Participants by Weight Category (>75 kg vs. ≤75 kg) [Count of Participants; unit: Participants]
  >75 kg | 55 | 55 | 110
  ≤75 kg | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Time-Concentration Curve From the Start of Dosing to 63 Days (AUC0-62) for Serum Pertuzumab
Description: For the analysis of AUC0-62days, participants in the Per Protocol Pharmacokinetics (PK) Analysis Population (PAP) with missing Day 63 PK pertuzumab concentration data or with a Day 63 PK sample time deviation outside a +/-120-hour window of planned sampling time were excluded. Participants were excluded from the PAP for the following reasons: 1. The participant violates inclusion or exclusion criteria regarding body mass index (BMI), use of prohibited medications and concomitant subcutaneous, intravenous (IV), or any parenteral drugs, participation in an investigational drug or device study, current chronic daily treatment with corticosteroids, and receipt of IV antibiotics for infection. 2. An SC injection site other than thigh is used; 3. Any participant whose injection is not successfully performed.
Time Frame: Predose (0 hour) and 2, 6, and 12 hours postdose on Day 1, and postdose on Days 2, 3, 5, 7, 9, 11, 15, 22, 35, 49, and 63
Population: Per Protocol PK Analysis Population for Pertuzumab AUC0-62 (PPAP1): includes all randomized participants who were treated and adhered to the pre-specified protocol criteria for general PK analysis and for pertuzumab AUC0-62 analysis specifically.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*day/mL
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 68 | 73
μg*day/mL | 1671.2 (27.5) | 1674.6 (23.2)
Statistical Analysis 1: Comparison: Arm 1: PH FDC SC Using a Handheld Syringe vs Arm 2: PH FDC SC Using the OBDS; Test type: Equivalence — The null hypothesis will be rejected and bioequivalence will be concluded if the bounds of the 90% CI for the geometric mean ratio of the AUC0-62 values for pertuzumab by administration using OBDS (Arm 2) relative to the handheld syringe (Arm 1) are entirely contained within standard bioequivalence margins (0.8 to 1.25); Geometric Mean Ratio (GMR) = 1.00, 90% CI 2-sided [0.93 to 1.08] — GMR of test treatment group (Arm 2: PH FDC SC using OBDS) to reference treatment group (Arm 1: PH FDC SC using handheld syringe)

2. Primary Outcome: Area Under the Time-Concentration Curve From the Start of Dosing to 63 Days (AUC0-62) for Serum Trastuzumab
Description: For the analysis of AUC0-62days, participants in the Per Protocol Pharmacokinetics (PK) Analysis Population (PAP) with missing Day 63 PK trastuzumab concentration data or with a Day 63 PK sample time deviation outside a +/-120-hour window of planned sampling time were excluded. Participants were excluded from the PAP for the following reasons: 1. The participant violates inclusion or exclusion criteria regarding body mass index (BMI), use of prohibited medications and concomitant subcutaneous, intravenous (IV), or any parenteral drugs, participation in an investigational drug or device study, current chronic daily treatment with corticosteroids, and receipt of IV antibiotics for infection. 2. An SC injection site other than thigh is used; 3. Any participant whose injection is not successfully performed.
Time Frame: as for outcome 1
Population: Per Protocol PK Analysis Population for Trastuzumab AUC0-62 (TPAP1): includes all randomized participants who were treated and adhered to the pre-specified protocol criteria for general PK analysis and for trastuzumab AUC0-62 analysis specifically.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*day/mL
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 68 | 73
μg*day/mL | 1341.2 (31.4) | 1347.1 (23.6)
Statistical Analysis 1: Comparison: Arm 1: PH FDC SC Using a Handheld Syringe vs Arm 2: PH FDC SC Using the OBDS; Test type: Equivalence — The null hypothesis will be rejected and bioequivalence will be concluded if the bounds of the 90% CI for the geometric mean ratio of the AUC0-62 values for trastuzumab by administration using OBDS (Arm 2) relative to the handheld syringe (Arm 1) are entirely contained within standard bioequivalence margins (0.8 to 1.25); Geometric Mean Ratio (GMR) = 1.00, 90% CI 2-sided [0.93 to 1.09] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Serum Concentration (Cmax) of Pertuzumab
Description: For analysis of Cmax, participants from the Per Protocol PK Analysis Population (PAP) with two or more missing PK pertuzumab concentration data on any of Days 3, 5, 7, 9 or 11 were excluded. Participants were excluded from the PAP for the following reasons: 1. The participant violates inclusion or exclusion criteria regarding body mass index (BMI), use of prohibited medications and concomitant subcutaneous, intravenous (IV), or any parenteral drugs, participation in an investigational drug or device study, current chronic daily treatment with corticosteroids, and receipt of IV antibiotics for infection. 2. An SC injection site other than thigh is used; 3. Any participant whose injection is not successfully performed.
Time Frame: as for outcome 1
Population: Per Protocol PK Analysis Population for Pertuzumab Cmax (PPAP2): includes all randomized participants who were treated and adhered to the pre-specified protocol criteria for general PK analysis and for pertuzumab Cmax analysis specifically.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per millilitre (μg/mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 68 | 74
microgram per millilitre (μg/mL) | 63.4 (32.2) | 65.8 (24.7)
Statistical Analysis 1: Comparison: Arm 1: PH FDC SC Using a Handheld Syringe vs Arm 2: PH FDC SC Using the OBDS; Test type: Equivalence — The null hypothesis will be rejected and bioequivalence will be concluded if the bounds of the 90% CI for the geometric mean ratio of the Cmax values for pertuzumab by administration using OBDS (Arm 2) relative to the handheld syringe (Arm 1) are entirely contained within standard bioequivalence margins (0.8 to 1.25); Geometric Mean Ratio (GMR) = 1.04, 90% CI 2-sided [0.96 to 1.12] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Maximum Serum Concentration (Cmax) of Trastuzumab
Description: For analysis of Cmax, participants from the Per Protocol PK Analysis Population (PAP) with two or more missing PK trastuzumab concentration data on any of Days 3, 5, 7, 9 or 11 were excluded. Participants were excluded from the PAP for the following reasons: 1. The participant violates inclusion or exclusion criteria regarding body mass index (BMI), use of prohibited medications and concomitant subcutaneous, intravenous (IV), or any parenteral drugs, participation in an investigational drug or device study, current chronic daily treatment with corticosteroids, and receipt of IV antibiotics for infection. 2. An SC injection site other than thigh is used; 3. Any participant whose injection is not successfully performed.
Time Frame: as for outcome 1
Population: Per Protocol PK Analysis Population for Trastuzumab Cmax (TPAP2): includes all randomized participants who were treated and adhered to the pre-specified protocol criteria for general PK analysis and for trastuzumab Cmax analysis specifically.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per millilitre (μg/mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 68 | 74
microgram per millilitre (μg/mL) | 59.8 (33.8) | 62.0 (25.2)
Statistical Analysis 1: Comparison: Arm 1: PH FDC SC Using a Handheld Syringe vs Arm 2: PH FDC SC Using the OBDS; Test type: Equivalence — The null hypothesis will be rejected and bioequivalence will be concluded if the bounds of the 90% CI for the geometric mean ratio of the Cmax values for trastuzumab by administration using OBDS (Arm 2) relative to the handheld syringe (Arm 1) are entirely contained within standard bioequivalence margins (0.8 to 1.25); Geometric Mean Ratio (GMR) = 1.04, 90% CI 2-sided [0.95 to 1.13] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Observed Serum Concentration of Pertuzumab on Day 22
Time Frame: Day 22
Population: The Per Protocol PK Population (PAP) includes all randomized participants who were treated and adhered to the pre-specified protocol criteria. Only participants who provided PK samples on Day 22 were included in this analysis.
Measure: Mean (Standard Deviation); unit: microgram per millilitre (μg/mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 69 | 73
microgram per millilitre (μg/mL) | 34.2 (10.6) | 34.6 (8.79)

6. Secondary Outcome: Observed Serum Concentration of Trastuzumab on Day 22
Time Frame: Day 22
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: microgram per millilitre (μg/mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 69 | 73
microgram per millilitre (μg/mL) | 29.9 (10.7) | 29.5 (6.72)

7. Secondary Outcome: Observed Serum Concentration of Pertuzumab on Day 63
Time Frame: Day 63
Population: The Per Protocol PK Population (PAP) includes all randomized participants who were treated and adhered to the pre-specified protocol criteria. Only participants who provided PK samples on Day 63 were included in this analysis.
Measure: Mean (Standard Deviation); unit: microgram per millilitre (μg/mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 69 | 74
microgram per millilitre (μg/mL) | 6.23 (3.64) | 6.23 (5.42)

8. Secondary Outcome: Observed Serum Concentration of Trastuzumab on Day 63
Time Frame: Day 63
Population: as for outcome 7
Measure: Median (Full Range); unit: microgram per millilitre (μg/mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 69 | 74
microgram per millilitre (μg/mL) | 1.00 [NA to 6.82] — The values for the majority of participant samples (n = 63) were lower than reportable (i.e., below the minimum quantifiable concentration of 1 ug/mL); thus, the lower limit of the full range could not be calculated. | 1.00 [NA to 35.2] — The values for the majority of participant samples (n = 55) were lower than reportable (i.e., below the minimum quantifiable concentration of 1 ug/mL); thus, the lower limit of the full range could not be calculated.

9. Secondary Outcome: Area Under the Time-Concentration Curve From the Start of Dosing Extrapolated to Infinity (AUC0-∞) for Serum Pertuzumab
Time Frame: as for outcome 1
Population: The Per Protocol PK Population (PAP) includes all randomized participants who were treated and adhered to the pre-specified protocol criteria. The number analyzed includes participants in the PAP with adequate concentration profiles, which allowed for individual PK parameters to be estimated.
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
μg*day/mL | 1930 (593) | 1860 (454)

10. Secondary Outcome: Area Under the Time-Concentration Curve From the Start of Dosing Extrapolated to Infinity (AUC0-∞) for Serum Trastuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
μg*day/mL | 1440 (453) | 1410 (331)

11. Secondary Outcome: Observed Time to Maximum Serum Concentration (Tmax) of Pertuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
Days | 4.00 [1.94 to 21.01] | 4.00 [1.99 to 21.02]

12. Secondary Outcome: Observed Time to Maximum Serum Concentration (Tmax) of Trastuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
Days | 4.01 [1.94 to 10.08] | 4.00 [1.99 to 13.91]

13. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Pertuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
Days | 15.6 [6.85 to 56.4] | 15.1 [7.86 to 24.6]

14. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Trastuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
Days | 8.93 [5.88 to 26.8] | 8.43 [5.89 to 19.0]

15. Secondary Outcome: Apparent Drug Clearance (CL/F) of Pertuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millilitres per day (mL/day)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
millilitres per day (mL/day) | 347 (124) | 361 (102)

16. Secondary Outcome: Apparent Drug Clearance (CL/F) of Trastuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millilitres per day (mL/day)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
millilitres per day (mL/day) | 469 (172) | 481 (122)

17. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Pertuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millilitres (mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
millilitres (mL) | 7670 (2030) | 7730 (2250)

18. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Trastuzumab
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: millilitres (mL)
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 70 | 74
millilitres (mL) | 6320 (2890) | 6030 (1980)

19. Secondary Outcome: Summary of the Number of Participants With at Least One Adverse Event, With Severity Determined According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0)
Description: The adverse event (AE) severity grading scale NCI CTCAE v5.0 was used for assessing AE severity. Any AEs for which the NCI CTCAE v5.0 did not provide a grading scale, the standard four-point scale from 1 to 4 (mild, moderate, severe, life-threatening) was used. The terms "severe" and "serious" are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs were counted only once per participant at the highest (worst) grade. AEs to monitor included administration-related reactions, hypersensitivity and anaphylaxis, diarrhoea, rash, cardiac dysfunction, neutropenia or febrile neutropenia, mucositis, and interstitial lung disease.
Time Frame: From study drug dose until safety follow-up visit (up to 7 months)
Population: Safety population: all participants who received the single dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
Participants
  Any Adverse Event (AE) | 70 | 71
  AE with Fatal Outcome | 0 | 0
  Serious AE | 1 | 0
  Related Serious AE | 0 | 0
  Grade 3 to 4 AE | 1 | 0
  AE Leading to Drug Interruption | 0 | 0
  Device Related AE | 0 | 0
  Any AE to Monitor | 63 | 59
  AE to Monitor: Anaphylaxis and Hypersensitivity, Any Grade | 48 | 36
  AE to Monitor: Anaphylaxis and Hypersensitivity, Grade ≥3 | 0 | 0
  AE to Monitor: Infusion/Admin. Related Reactions Within 24 hours, Any Grade | 62 | 55
  AE to Monitor: Infusion/Admin. Related Reactions Within 24 hours, Grade ≥3 | 0 | 0
  AE to Monitor: Rash/Skin Reactions, Any Grade | 0 | 0
  AE to Monitor: Diarrhoea, Any Grade | 17 | 9
  AE to Monitor: Diarrhoea, Grade ≥3 | 0 | 0
  AE to Monitor: Cardiac Dysfunction, Any Grade | 0 | 0
  AE to Monitor: Interstitial Lung Disease, Any Grade | 0 | 0
  AE to Monitor: Neutropenia/Febrile Neutropenia, Any Grade | 0 | 1
  AE to Monitor: Neutropenia/Febrile Neutropenia, Grade ≥3 | 0 | 0
  AE to Monitor: Serious Mucositis, Any Grade | 0 | 0

20. Secondary Outcome: Change From Baseline Left Ventricular Ejection Fraction (LVEF) Over Time
Description: Echocardiography was used to assess left ventricular ejection fraction (LVEF) values. The screening LVEF assessment had to be performed within ≤28 days prior to randomization and the LVEF value must have been ≥55% to be eligible for the study.
Time Frame: Baseline, once between Days 20 and 35, and once between Days 56 and 63
Population: Safety population: all participants who received the single dose of study treatment. The number analyzed represents all participants with available data at a given timepoint.
Measure: Mean (Standard Deviation); unit: Percentage points of LVEF
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
Percentage points of LVEF
  Baseline (BL) - Value at Visit | 61.55 (3.56) | 60.99 (3.82)
  Change from BL - Day 20 to 35: number analyzed (Participants) | 69 | 74
  Change from BL - Day 20 to 35 | 0.10 (4.88) | -0.94 (4.06)
  Change from BL - Day 56 to 63: number analyzed (Participants) | 69 | 73
  Change from BL - Day 56 to 63 | -0.87 (5.04) | -0.20 (4.29)
  Change from BL - Minimum Value at Anytime | -2.09 (4.39) | -2.36 (3.84)
  Change from BL - Maximum Value at Anytime | 1.32 (5.01) | 1.23 (3.70)

21. Secondary Outcome: Change From Baseline Pulse Rate Over Time
Description: Vital sign measurements were taken after the participant had remained resting in a semi-supine position for at least 5 minutes. The minimum and maximum values are, respectively, the smallest and largest values obtained at any point after baseline, including any repeat and unscheduled measurements.
Time Frame: Baseline, Days 2, 7, 22, and 63
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
beats per minute
  Baseline (BL) - Value at Visit | 58.24 (9.30) | 59.30 (10.89)
  Change from BL at Day 2 | 7.04 (8.51) | 6.51 (10.86)
  Change from BL at Day 7: number analyzed (Participants) | 69 | 73
  Change from BL at Day 7 | 1.80 (8.63) | 4.34 (11.39)
  Change from BL at Day 22: number analyzed (Participants) | 70 | 73
  Change from BL at Day 22 | 5.40 (11.52) | 5.14 (11.91)
  Change from BL at Day 63: number analyzed (Participants) | 70 | 74
  Change from BL at Day 63 | 2.47 (8.64) | 4.16 (10.87)
  Change from BL - Minimum Value at Anytime | -2.49 (7.67) | -1.78 (9.17)
  Change from BL - Maximum Value at Anytime | 14.79 (15.06) | 13.19 (12.09)

22. Secondary Outcome: Change From Baseline Respiratory Rate Over Time
Description: as for outcome 21
Time Frame: Baseline, Days 2, 7, 22, and 63
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
breaths per minute
  Baseline (BL) - Value at Visit | 15.71 (1.61) | 15.50 (1.49)
  Change from BL at Day 2 | -0.22 (2.22) | -0.03 (2.39)
  Change from BL at Day 7: number analyzed (Participants) | 69 | 73
  Change from BL at Day 7 | 0.00 (2.31) | 0.04 (2.10)
  Change from BL at Day 22: number analyzed (Participants) | 70 | 73
  Change from BL at Day 22 | -0.34 (1.68) | 0.53 (2.04)
  Change from BL at Day 63: number analyzed (Participants) | 69 | 74
  Change from BL at Day 63 | -0.19 (2.30) | 0.15 (2.61)
  Change from BL - Minimum Value at Anytime | -1.86 (1.69) | -1.64 (2.00)
  Change from BL - Maximum Value at Anytime | 1.44 (1.96) | 1.93 (2.08)

23. Secondary Outcome: Change From Baseline Systolic Blood Pressure Over Time
Description: as for outcome 21
Time Frame: Baseline, Days 2, 7, 22, and 63
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
beats per minute
  Baseline (BL) - Value at Visit | 118.33 (9.19) | 116.09 (9.68)
  Change from BL at Day 2 | -1.44 (7.90) | 0.61 (9.02)
  Change from BL at Day 7: number analyzed (Participants) | 69 | 73
  Change from BL at Day 7 | 4.55 (7.14) | 4.99 (9.20)
  Change from BL at Day 22: number analyzed (Participants) | 70 | 73
  Change from BL at Day 22 | 3.60 (10.76) | 5.23 (10.70)
  Change from BL at Day 63: number analyzed (Participants) | 70 | 74
  Change from BL at Day 63 | 4.70 (9.51) | 5.53 (9.64)
  Change from BL - Minimum Value at Anytime | -4.68 (7.97) | -3.51 (8.00)
  Change from BL - Maximum Value at Anytime | 11.17 (9.96) | 12.78 (11.13)

24. Secondary Outcome: Change From Baseline Diastolic Blood Pressure Over Time
Description: as for outcome 21
Time Frame: Baseline, Days 2, 7, 22, and 63
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
beats per minute
  Baseline (BL) - Value at Visit | 70.50 (7.55) | 70.38 (7.20)
  Change from BL at Day 2 | -1.99 (6.86) | -2.12 (6.49)
  Change from BL at Day 7: number analyzed (Participants) | 68 | 73
  Change from BL at Day 7 | 3.04 (6.82) | 2.62 (7.04)
  Change from BL at Day 22: number analyzed (Participants) | 70 | 73
  Change from BL at Day 22 | 3.43 (7.13) | 4.16 (7.67)
  Change from BL at Day 63: number analyzed (Participants) | 70 | 74
  Change from BL at Day 63 | 3.96 (7.86) | 3.64 (8.36)
  Change from BL - Minimum Value at Anytime | -4.58 (7.16) | -4.30 (6.13)
  Change from BL - Maximum Value at Anytime | 8.13 (7.11) | 8.65 (7.13)

25. Secondary Outcome: Number of Participants With Normal or Abnormal Electrocardiogram Results at Baseline and Post-Baseline Anytime, as Determined by the Investigator
Description: For safety monitoring purposes, the investigator was required to review, sign, and date all electrocardiogram (ECG) reports. Any morphologic waveform changes or other ECG abnormalities were documented by the investigator. Post-baseline, if all examinations were normal, then it was categorized as 'Normal'. If any abnormality was reported, then it was categorized as 'Abnormal'. 'Clinically significant' is a subset of the abnormal category.
Time Frame: At Baseline (predose) and Post-Baseline (postdose Days 2, 7, 22, and 63)
Population: Safety population: all participants who received the single dose of study treatment. The number analyzed represents all participants with available data at baseline and at least at one post-baseline timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
Participants
  Baseline: Normal ECG | 48 | 42
  Baseline: Abnormal ECG | 24 | 32
  Baseline: Abnormal and Clinically Significant ECG | 0 | 0
  Post-Baseline: Normal ECG | 42 | 35
  Post-Baseline: Abnormal ECG | 30 | 39
  Post-Baseline: Abnormal and Clinically Significant ECG | 0 | 0

26. Secondary Outcome: Number of Participants With Adverse Events Based on Laboratory Test Abnormalities
Description: Not every laboratory abnormality qualified as an adverse event. A laboratory test result had to be reported as an adverse event if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; was clinically significant in the investigator's judgment.
Time Frame: From Baseline until Day 63
Population: Safety population: all participants who received the single dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
Participants
  Alanine aminotransferase increased | 0 | 1
  Hepatic enzyme increased | 0 | 1
  Transaminases increased | 1 | 0
  Anaemia | 0 | 1
  Neutropenia | 0 | 1

27. Secondary Outcome: Pain Score at the Injection Site, Assessed by the Participant Using the 100-millimetre (mm) Visual Analog Scale
Description: Pain intensity scores were assessed by the participants using the Visual Analog Scale (VAS) on a line measuring between 0 mm ('no pain') and 100 mm ('unbearable pain'). The VAS was completed in both study arms to assess the level of pain experienced by the participant in relation to the injection of Phesgo. On Day 1, pain assessments were performed prior to, during, and immediately after injection of Phesgo when the needle or device was removed, and 2 hours after injection.
Time Frame: Day 1: pre-dose, during drug injection, after drug injection while removing the device or syringe, and 2 hours after drug injection
Population: Safety population: all participants who received the single dose of study treatment. The number analyzed indicates all participants who responded to the questionnaire at a given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 72 | 74
score on a scale
  Prior to Injection | 0.68 (1.45) | 0.50 (1.52)
  During Injection | 6.85 (8.79) | 8.95 (10.28)
  Immediately Post-Injection | 8.56 (12.62) | 5.04 (7.82)
  2 Hours After Injection | 3.11 (5.29) | 1.62 (5.97)

28. Secondary Outcome: Number of Participants With Skin Irritation and Sensitization Reactions at the Injection Site, as Reported by Investigators in the Device Monitoring Questionnaire
Description: Skin irritation and sensitization reactions at the site of injection caused by the adhesion of the OBDS to the skin were assessed by the study staff using the device monitoring questionnaire in the eCRF. Dermal effects were reported on a scale from 0 (no evidence or irritation) to 7 (strong reaction spreading beyond test site). Other effects were reported on a separate scale from 0 (no evidence) to 7 (small petechial eruptions or scabs).
Time Frame: Prior to injection and after injection on Day 1
Population: The analysis only included healthcare professionals that treated participants in Arm 2: PH FDC SC Using OBDS who received the single dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 74
Participants
  Prior to Injection, Dermal Effects: 0 - No Evidence or Irritation | 74
  After Injection, Dermal Effects: 0 - No Evidence or Irritation | 62
  After Injection, Dermal Effects: 1 - Minimal Erythema | 12
  Prior to Injection, Other Effects: 0 - No Evidence or Irritation | 74
  After Injection, Other Effects: 0 - No Evidence or Irritation | 73
  After Injection, Other Effects: 1 - Slight Glazed Appearance | 1

29. Secondary Outcome: Number of Participants by Their Ratings of the Comfort of Wearing the On-Body Delivery System Device, as Reported in the Device Monitoring Questionnaire
Description: Participants in the Phesgo OBDS arm completed the device monitoring questionnaire the injection with the OBDS. The questionnaire assessed the following criteria: ease of device attachment, attachment during the injection, ease of device removal, and overall wearing comfort, which were each rated on a three-point scale as "Good", "Acceptable", or "Poor".
Time Frame: Day 1
Population: The analysis only included participants in Arm 2: PH FDC SC Using OBDS who received the single dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 74
Participants
  Ease of Device Attachment: Good | 74
  Ease of Device Attachment: Acceptable | 0
  Ease of Device Attachment: Poor | 0
  Attachment of Device During Injection: Good | 73
  Attachment of Device During Injection: Acceptable | 1
  Attachment of Device During Injection: Poor | 0
  Ease of Device Removal: Good | 67
  Ease of Device Removal: Acceptable | 6
  Ease of Device Removal: Poor | 1
  Overall Wearing Comfort: Good | 67
  Overall Wearing Comfort: Acceptable | 7
  Overall Wearing Comfort: Poor | 0

30. Secondary Outcome: Number of Healthcare Professionals by Their Responses to the Device Monitoring Questionnaire Regarding Use of the On-Body Delivery System Device
Description: Details of performance and ease of use of the on-body delivery system (OBDS) were reported by site staff, using the device monitoring questionnaire in the eCRF. This included the following: Preparation of the injection site, Preparation of the OBDS, Prefilled cartridge inspection before insertion in the OBDS, Positioning and attachment of the OBDS on the anterior thigh, Drug delivery, and OBDS administration failures.
Time Frame: Day 1
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2: PH FDC SC Using the OBDS
Number analyzed (Participants) | 74
Participants
  Was the Injection Site Prepared as per Protocol?: Yes | 74
  Was the Injection Site Prepared as per Protocol?: No | 0
  Was the Injection Device Prepared as per Protocol?: Yes | 74
  Was the Injection Device Prepared as per Protocol?: No | 0
  Was the Body Positioning of the Device Compliant with Protocol?: Yes | 74
  Was the Body Positioning of the Device Compliant with Protocol?: No | 0
  Were There any Findings from the Cartridge Inspection?: Yes | 0
  Were There any Findings from the Cartridge Inspection?: No | 74
  Were There any Issues with the Attachment of the Device to the Body?: Yes | 0
  Were There any Issues with the Attachment of the Device to the Body?: No | 74
  Did you Experience any Device Failure?: Yes | 0
  Did you Experience any Device Failure?: No | 74
  Has Needle Been Inserted?: Yes | 74
  Has Needle Been Inserted?: No | 0
  Has Another Device Been Used?: Yes | 0
  Has Another Device Been Used?: No | 74

ADVERSE EVENTS:
Time Frame: From study drug dose until safety follow-up visit (up to 7 months)
Description: All adverse events were to be reported until Day 63 after the single dose of study drug. After this point only death, serious adverse events, adverse events, or adverse event of special interest that were related to study drug were reported until the 7-month safety follow-up visit.
Arm/Group | Arm 1: PH FDC SC Using a Handheld Syringe | Arm 2: PH FDC SC Using the OBDS
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/74
Other Adverse Events (participants affected / at risk) | 70/72 | 69/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: PH FDC SC Using a Handheld Syringe (N=72) | Arm 2: PH FDC SC Using the OBDS (N=74)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: PH FDC SC Using a Handheld Syringe (N=72) | Arm 2: PH FDC SC Using the OBDS (N=74)
Injection related reaction (Injury, poisoning and procedural complications) | 48 (48) | 36 (36)
Injection site reaction (General disorders) | 17 (17) | 18 (19)
Fatigue (General disorders) | 4 (4) | 6 (6)
Injection site bruising (General disorders) | 3 (3) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 12 (13) | 15 (15)
COVID-19 (Infections and infestations) | 6 (6) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 9 (9)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 18 (21) | 17 (19)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 (8) | 8 (8)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Seasonal allergy (Immune system disorders) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT05275010/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT05275010/SAP_001.pdf